CLINICAL TRIAL: NCT04834440
Title: Ropivacaine Use in Femoral Nerve Block; What is the Minimal Effective Analgesic Concentration (MEAC 90)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Healthpoint Hospital (Other)
Responsible Party: Principal Investigator, Ahmad Muhammad Taha, Consultant of anesthesia, Healthpoint Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MF2467-2021-14
Record Dates: First submitted 2021-03-31; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Ropivacaine — all patients will receive femoral nerve block using same volume of ropivacaine but in different concentrations

SUMMARY:
The aim of this study is to determine the minimal effective ropivacaine concentration required to provide adequate analgesic femoral nerve block in 90% of patients (MEAC90)

DETAILED DESCRIPTION:
* Before induction of GA, all patients will receive sciatic, obturator, lateral femoral cutaneous and femoral nerve blocks.
* The femoral nerve block will be performed using 15ml of ropivacaine which concentration relied on the response of the previous patient.
* Based on biased-coin design up-down sequential method: when a patient has a negative response, the next patient will receive a concentration 0.01% w/v higher. However if he has a positive response, the next patient will be randomized to receive either the same ropivacaine concentration or a concentration 0.01% w/v less.
* Patients with pain free recovery will be considered to have positive response.
* Patients' responses will be analyzed to calculate the MEAC90

ELIGIBILITY:
Inclusion Criteria:

* Patients, who are scheduled for knee ligament reconstruction

Exclusion Criteria:

* <18 y,
* ASA physical class greater >III

  * BMI >40 has any contraindication for medications or techniques used in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
effective analgesic femoral nerve block | in recovery unit (one hour after surgery)
  postoperative pain. it will be assessed using numerical rating scale (NRS). NRS, 0 = no pain; 10 = worst pain imaginable; if NRS ≥ 3, pain (ineffective block) is considered, other wise a successful block will be considered.

CONTACTS AND LOCATIONS:
Locations (1):
- Healthpoint Hospital, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No